CLINICAL TRIAL: NCT00936637
Title: A 16-Week Growth Study of an Extensively Hydrolyzed Infant Formula, 3 Months Treatment and 1 Month Follow-up for a Duration of 4 Months.
Brief Title: Effects on Growth of an Extensively Hydrolyzed Formula Fed to Term
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Perrigo Nutritionals (Industry)
Responsible Party: Cynthia Barber, PhD; Vice President of Regulatory, Medical and Clinical Affairs, PBM Products
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: UVA Growth Study
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Growth

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- Extensively hydrolyzed infant formula (Experimental)
  Interventions: Other: Extensively hydrolyzed infant formula

INTERVENTIONS:
Other: Extensively hydrolyzed infant formula

SUMMARY:
The purpose of this study is to assess growth in infants who are fed an extensively hydrolyzed formula.

ELIGIBILITY:
Inclusion Criteria:

* At birth:

  * Healthy, term (37-42 weeks) infant
  * Weight for length between the 10th and 90th percentile according to the National Center for Health Statistics (NCHS) growth charts
* At time of enrollment:

  * < or = 21 days post-natal age
  * Weight for length between the 10th and 90th percentile according to the National Center for Health Statistics (NCHS) growth charts
  * Exclusively formula fed
  * Written informed consent of parent/guardian

Exclusion Criteria:

* At the time of enrollment: partially human-milk fed; fed baby/solid foods
* Conditions requiring feedings other than those specified in the protocol
* Documented or suspected cow's milk allergy and/or soy protein allergies
* Major congenital deformities
* Suspected or documented systemic or congenital infections
* Evidence of cardiac, respiratory, hematological, gastrointestinal, or other systemic diseases
* Participation in any other clinical trial

Ages: 1 Day to 21 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
An extensively hydrolyzed formula is nutritionally adequate for normal growth of healthy full-term infants | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia M Barber, PhD, Study Director — Perrigo Nutritionals
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States